CLINICAL TRIAL: NCT02596347
Title: The Role of JAK2 in Alveolar Macrophages in Chronic Beryllium Disease
Brief Title: The Role of JAK2 in Alveolar Macrophages (AM's) in Chronic Beryllium Disease (CBD)
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Li Li, Dr., National Jewish Health
Other Study IDs: 2877
Record Dates: First submitted 2015-10-29; First posted 2015-11-04 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Chronic Beryllium Disease (CBD); Beryllium Sensitization (BeS)
MeSH Terms: interventions — Blood Specimen Collection; Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid 4 heparin tubes for PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Beryllium Sensitization (BeS): Blood draw
  Interventions: Procedure: Blood draw
- Chronic Beryllium Disease(CBD): blood draw BAL
  Interventions: Procedure: Blood draw; Procedure: bronchoscopy

INTERVENTIONS:
Procedure: Blood draw — We will draw 4 heparin tubes for peripheral blood mononuclear cells (PBMC)
Procedure: bronchoscopy — CBD subjects will undergo a bronchoscopy with lavage. This is the passage of a think flexible tube through the nose into the windpipe then into the bronchial tubes. Sterile saltwater solution is through the flexible tube then immediately removed.
  Other Names: BAL
  Groups: Chronic Beryllium Disease(CBD)

SUMMARY:
Current studies suggest that alveolar macrophages (AM) act as silencers of most immune responses in the lung. However, in pathological conditions, such as asthma, hypersensitivity pneumonitis, and sarcoidosis, AMs become involved in the maintenance and further expansion of the immune response in the target organ. The Investigator has preliminary data demonstrating that CBD AMs at the site of disease involvement (bronchoalveolar lavage, BAL) display an activated cell surface phenotype compared to AMs from healthy controls. Furthermore, exciting data from our group demonstrates significant differences in gene expression profiles between CBD and Beryllium Sensitivity (BeS) bronchial alveolar lavage (BAL) cells, in pivotal immune response genes and networks. Specifically, the Investigator has found the JAK/STAT pathway and the JAK2 gene was dramatically overexpressed in CBD BAL cells. In addition, constitutively phosphorylated JAK2 (pJAK2) was found in AMs from Chronic Beryllium Disease (CBD) patients by Westernblot and was increased after beryllium (Be) stimulation for 30 min. Moreover, the JAK2 inhibitor TG101348 significantly inhibited Be-induced CBD AMs TNFa and IFNy production. Meanwhile, overexpression of the JAK2 inhibitor SOCS 1 (suppressors of cytokine signaling) protein decreased Be-induced TNFa production from AMs. Based on this information, the Investigator hypothesizes that CBD AMs overexpress JAK2, which augments the immune response to Be and development of CBD but not BeS.

The investigators believe that these studies are highly innovative since they will undoubtedly shed light on exposure-mediated immune dysregulation in Alveolar Macrophages (AMs) that lead to disease development and likely progression and with additional study of this pathway will reveal potential biomarkers for clinical prognosis and diagnosis. The results obtained from this study will improve the investigators understanding of factors involved in the development of Chronic Beryllium disease (CBD), as well as define targets for therapy, and will serve as a model of other exposure-related immune responses and environmentally-induced chronic diseases. Most importantly, these studies will provide the investigator with preliminary data to submit a high quality R01, allowing the Investigator to apply similar approaches to other genes, define a potential target for this and other similar immune-mediated diseases and continue research efforts at National Jewish Health (NJH.)

ELIGIBILITY:
Inclusion Criteria:

* Chronic Beryllium Disease - These individuals will meet the following inclusion criteria:

Inclusion Criteria:

1. History of beryllium exposure;
2. Positive blood and/or bronchoalveolar lavage (BAL) Beryllium Lymphocyte Proliferation Tests (BeLPT);
3. Biopsy-proven pathologic changes consistent with CBD, specifically non-caseating granulomas and/or mononuclear cell interstitial infiltrates .

Beryllium Sensitization - These individuals will meet the following inclusion criteria:

Inclusion Criteria:

1. History of beryllium exposure;
2. Two or more positive blood beryllium lymphocyte proliferation tests (BeLPT) or positive bronchoalveolar lavage (BAL) BeLPT;
3. Normal lung tissue (no histology suggestive of CBD).

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those diagnosed with Beryllium Sensitization. Those diagnosed with Chronic beryllium disease
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-04; Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome for the aims is the downregulation of Th1 cytokine TNFalpha with the inhibition of the JAK2 using siRNA and the inhibitor INCB018424, CEP-701 and TG101348 in CBD or overexpression of the JAK2 gene. | year 1
  As the primary outcome is the downregulation of TNFalpha level with the inhibition of the JAK2 using the inhibitor TG101348 in CBD, we expect a 50% reduction with a standard deviation of 0.2 based on our preliminary data. We will have more than 95% power with n=6 CBD patients for these aims.
The secondary outcomes for the aims are the changes in BeLPT and AMs phenotype from BeS, CBD and Healthy controls (HC). | year 2
  The investigator will use repeated measure Welch's ANOVA in SAS 9.4, which correctly accounts for the correlation between measurements and allows for comparisons within and between groups. Normalizing transformations will be performed when necessary to conform to model assumptions and Mauchly's sphericity test will be assessed and adjustments will be added to the analysis as necessary. Estimate and contrast statements will be developed to test hypotheses of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Li L, Schmitt A, Reinhardt P, Greiner J, Ringhoffer M, Vaida B, Bommer M, Vollmer M, Wiesneth M, Dohner H, Schmitt M. Reconstitution of CD40 and CD80 in dendritic cells generated from blasts of patients with acute myeloid leukemia. Cancer Immun. 2003 Jul 16;3:8. PMID 12862419
- [Background] Greiner J, Ringhoffer M, Taniguchi M, Li L, Schmitt A, Shiku H, Dohner H, Schmitt M. mRNA expression of leukemia-associated antigens in patients with acute myeloid leukemia for the development of specific immunotherapies. Int J Cancer. 2004 Feb 20;108(5):704-11. doi: 10.1002/ijc.11623. PMID 14696097
- [Background] Li L, Reinhardt P, Schmitt A, Barth TF, Greiner J, Ringhoffer M, Dohner H, Wiesneth M, Schmitt M. Dendritic cells generated from acute myeloid leukemia (AML) blasts maintain the expression of immunogenic leukemia associated antigens. Cancer Immunol Immunother. 2005 Jul;54(7):685-93. doi: 10.1007/s00262-004-0631-8. Epub 2004 Dec 31. PMID 15627212
- [Background] Greiner J, Li L, Ringhoffer M, Barth TF, Giannopoulos K, Guillaume P, Ritter G, Wiesneth M, Dohner H, Schmitt M. Identification and characterization of epitopes of the receptor for hyaluronic acid-mediated motility (RHAMM/CD168) recognized by CD8+ T cells of HLA-A2-positive patients with acute myeloid leukemia. Blood. 2005 Aug 1;106(3):938-45. doi: 10.1182/blood-2004-12-4787. Epub 2005 Apr 12. PMID 15827130
- [Background] Li L, Giannopoulos K, Reinhardt P, Tabarkiewicz J, Schmitt A, Greiner J, Rolinski J, Hus I, Dmoszynska A, Wiesneth M, Schmitt M. Immunotherapy for patients with acute myeloid leukemia using autologous dendritic cells generated from leukemic blasts. Int J Oncol. 2006 Apr;28(4):855-61. PMID 16525634
- [Background] Li Q, Li L, Shi W, Jiang X, Xu Y, Gong F, Zhou M, Edwards CK 3rd, Li Z. Mechanism of action differences in the antitumor effects of transmembrane and secretory tumor necrosis factor-alpha in vitro and in vivo. Cancer Immunol Immunother. 2006 Dec;55(12):1470-9. doi: 10.1007/s00262-006-0150-x. Epub 2006 Mar 23. PMID 16555058
- [Background] Giannopoulos K, Li L, Bojarska-Junak A, Rolinski J, Dmoszynska A, Hus I, Greiner J, Renner C, Dohner H, Schmitt M. Expression of RHAMM/CD168 and other tumor-associated antigens in patients with B-cell chronic lymphocytic leukemia. Int J Oncol. 2006 Jul;29(1):95-103. PMID 16773189
- [Background] Greiner J, Schmitt M, Li L, Giannopoulos K, Bosch K, Schmitt A, Dohner K, Schlenk RF, Pollack JR, Dohner H, Bullinger L. Expression of tumor-associated antigens in acute myeloid leukemia: Implications for specific immunotherapeutic approaches. Blood. 2006 Dec 15;108(13):4109-17. doi: 10.1182/blood-2006-01-023127. Epub 2006 Aug 24. PMID 16931630
- [Background] Schmitt M, Li L, Giannopoulos K, Chen J, Brunner C, Barth T, Schmitt A, Wiesneth M, Dohner K, Dohner H, Greiner J. Chronic myeloid leukemia cells express tumor-associated antigens eliciting specific CD8+ T-cell responses and are lacking costimulatory molecules. Exp Hematol. 2006 Dec;34(12):1709-19. doi: 10.1016/j.exphem.2006.07.009. PMID 17157168